CLINICAL TRIAL: NCT06288074
Title: Diagnosis and Treatment Strategy Optimization of Severe Pneumonia Based on Multi-omics Data Integration
Status: Recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Zhaohui Tong, Clinical Professor, Capital Medical University
Other Study IDs: SF-2022-1-1061
Record Dates: First submitted 2024-01-03; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Severe Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe community-acquired pneumonia
  Interventions: Diagnostic Test: Multi-omics tests
- Non-Severe community-acquired pneumonia
  Interventions: Diagnostic Test: Multi-omics tests
- Healthy control
  Interventions: Diagnostic Test: Multi-omics tests

INTERVENTIONS:
Diagnostic Test: Multi-omics tests — Biological sample collection for Multi-omics tests

SUMMARY:
Severe community-acquired pneumonia still has a high incidence and mortality, but the molecular mechanism and prognostic biomarkers of severe community-acquired pneumonia caused by different pathogens are still unclear, and the best treatment strategy has not been determined. Based on this, this project intends to take patients with severe community-acquired pneumonia caused by different pathogens as the research object, explore the molecular mechanism of severe community-acquired pneumonia from multiple angles, integrate relevant research data to evaluate the rationality of initial empirical medication, and lay the foundation for precise treatment of severe pneumonia. The research results will help to develop a new rapid and accurate target for clinical diagnosis and efficacy evaluation of severe pneumonia, and build a precise treatment system for severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

Age> 18 years old

Clinical diagnosis of community-acquired pneumonia

Exclusion Criteria:

Pregnancy, perinatal and lactating women

Combined immunosuppressive diseases: such as HIV, solid organ transplantation, solid organ/hematologic malignant tumor chemotherapy, rheumatic diseases or glomerular diseases need to take hormone/immunosuppressant therapy

Combined blood system diseases: such as leukemia reactions, aplastic anemia, neutropenia or deficiency of granulocytes, previous bone marrow/stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A prospective cohort including 100 patients with severe and 100 patients with non-severe community-acquired pneumonia and 100 healthy people was selected.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality | during hospitalization (up to day 14)

SECONDARY OUTCOMES:
Cause of death | during hospitalization (up to day 14)
Length of stay | during hospitalization (up to day 14)
Length of ICU stay | during hospitalization (up to day 14)
Expense during hospitalization | during hospitalization (up to day 14)
  All expenses incurred in hospitalization, including bed fee, examination fee, operation or treatment fee.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Institute of Respiratory Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD is to be uploaded to the public platform and made public to all researchers.